CLINICAL TRIAL: NCT00756379
Title: Randomized Trial of Comprehensive Lifestyle Modifications, Optimal Pharmacological Treatment and PET Imaging for Detection and Management of Stable Coronary Artery Disease
Brief Title: Century Trial, a Randomized Lifestyle Modification Study for Management of Stable Coronary Artery Disease
Acronym: Century
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, K.Lance Gould, Professor, Internal Medicine, Cardiology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-MS-08-0312
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular Disease; Atherosclerosis; Coronary Artery Disease; Coronary Stenosis
Keywords: Cardiovascular disease; Atherosclerosis; Coronary artery disease; Coronary perfusion defect; Absolute coronary flow; Lifestyle management; Cardiovascular rehabilitation; Cardiovascular dietary guidelines
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Coronary Artery Disease; Coronary Stenosis | interventions — JCAD protein, mouse

STUDY DESIGN:
Intervention Model Description: Study Intervention: PET diagnostic imaging offered in addition to current standard of care for the detection of coronary atherosclerosis.
  Comprehensive program of atherosclerotic risk factor modification, involving treatment to target lipid levels, blood pressure and diabetes control, smoking cessation, very low fat diet and aerobic exercise program.
  This is addition to standard current medical therapy as provided by primary referring physician. No experimental medication or procedure will be used. Clinic visits for patients education and consulting in the comprehensive program will be performed five times during the first year and semiannually thereafter.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive lifestyle modification (Experimental): P.E.T. guided comprehensive therapy program. The study intervention is Comprehensive therapy program for risk factor modification. The Comprehensive program of atherosclerotic risk factor modification involves treatment to target lipid levels, blood pressure and diabetes control, smoking cessation, very low fat diet and aerobic exercise program. This is in addition to standard current medical therapy as provided by primary physician. No experimental medications or procedures will be used.
  Interventions: Other: Comprehensive therapy program for risk factor modification
- Current standard of care (No Intervention): Current standard of care medical management as provided by primary physician.

INTERVENTIONS:
Other: Comprehensive therapy program for risk factor modification — Patients enrolled in the comprehensive therapy arm will have a baseline myocardial perfusion PET and the support of a team of professionals aiming to modify and minimize all the known CAD risk factors. During the 5 year follow-up they will be educated and guided toward a healthy lifestyle by a dietician, an exercise physiologist/cardiovascular physician specialist.
  Other Names: Coronary artery disease; Lifestyle management; Atherosclerosis; Cardiovascular disease management; Cardiovascular disease reversal
  Arms: Intensive lifestyle modification

SUMMARY:
The Century Trial is a single center Phase III randomized study sponsored by the Albert Weatherhead III Foundation and conducted by Dr. K. Lance Gould. The study hypothesis is that a combined image-treatment regimen of PET + comprehensive program of lifestyle modification and lipid lowering drugs to target lipid level will result in an improved cardiovascular risk score when compared to current standard optimal medical therapy, potentially resulting in a lower rate of death, non-fatal myocardial infarction (MI) and revascularization procedures during long term follow-up when compared with current standard of care. If our hypothesis is correct, we will not only improve our ability to prevent and treat CAD but we will also illustrate that, even with the expenses of behavioral interventions and imaging techniques, we can be very cost effective. This information may help patients at risk or with known CAD to obtain insurance coverage to prevent the disease as well as providing a more effective way of treating it.

DETAILED DESCRIPTION:
Advances in diagnostic imaging with expensive technologies and reimbursement policies that favor illness intervention rather than primary and secondary prevention have resulted in rising costs of health care and more people being deprived of its benefits (Sultz 2004, Bodenheimer 2002).

In the field of coronary artery disease (CAD) are several non-invasive imaging techniques for diagnostic and risk stratification purposes such as echocardiography, perfusion imaging (cardiac stress SPECT - single photon emission computed tomography - and stress PET - positron emission tomography), non-invasive cardiac computed tomography angiography (CTA) and combined perfusion-anatomy (PET-CT) studies. There are an estimated 40 million noninvasive cardiac tests performed each year (Mark DB 2003). For echocardiography and SPECT imaging, reimbursement from Medicare encompasses approximately 30% of all payments, totaling over $1 billion in the year 2000 (ACC 2003). There are, however, basic questions about cardiovascular imaging techniques that need to be addressed: how does technology benefit the patient? It is worth the cost? Is treatment plan enhanced? Is outcome better? Data are necessary for addressing these questions and if appropriate for acceptance among practicing physicians, patients and third party insurers.

The relevance of the proposed study, the CENTURY trial, lies in its original design, testing the impact of stress perfusion imaging by PET coupled with two different intensities of clinical management strategies (standard or comprehensive respectively). This study will examine post-test resource utilization and reduction of cardiovascular risk in patients with known disease or at high risk for CAD.

There will be a total of 1300 men and women enrolled with approximately 650 subjects randomized to one of two treatment arms. Eligible patients must have clinical indications for stress perfusion testing.

Following confirmation of eligibility and provision of signed informed consent, patients will be randomized to one of the two possible treatment strategies. At time of randomization patients will be assigned to "PET guided + comprehensive" versus "standard medical treatment."

Patients of both groups will have a baseline myocardial PET perfusion study to quantify the blood flow to the heart muscle, an electrocardiogram, an exercise treadmill stress test to assess exercise tolerance (fitness), a thorough review of the quality of their diet and a complete blood work covering individual lipid profiles. These tests and assessments will be repeated at 2 years and at 5 years.

In addition, subjects assigned to the standard medical management arm will be managed by current standard care provided by their primary referring physician and will be asked to come for clinic study visits annually for 5 years to document their medical and lifestyle management. The PET scan results will be blinded until the end of the study to the standard of care management group.

Subjects enrolled in the comprehensive medical management arm will have the support of a team of professionals focusing on atherosclerotic risk factor modification that involves recommended treatment to target lipid levels, blood pressure and diabetes control, smoking cessation, very low fat diet and aerobic exercise program. This is in addition to standard current medical therapy as provided by the primary referring physician.

No experimental medication or procedures will be used. Clinic visits for subject's education and consulting in the comprehensive program will be performed five times during the first year and semiannually thereafter.

At the end of the first 5 years, patients in the "comprehensive" medical management arm will be offered an additional 5-year follow-up at the current study location once a year.

The extended follow-up on cardiovascular or other adverse events for the "current standard of care" group will be based on yearly telephone or mail follow-up.

Both groups will have a full consultation visit, exercise treadmill and dipyridamole PET scan at the end of the total 10 years follow-up, replicating the current initial 5-year follow-up visit protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be competent to provide written informed consent.
* Subjects must sign an Institutional Review Board (IRB) approved Informed Consent Form (ICF) and HIPAA Authorization prior to the initiation of any study procedures.
* Men and women age ≥40

  _ Indication for stress perfusion testing
* Appropriate Indications for stress perfusion testing:
* Suspected CAD:
* Men with any chest pain syndrome and two other risk factors
* Women >50 years old with any chest pain syndrome and two other risk factors
* Asymptomatic men and women >50 years with at least three other risk factors* or Coronary Calcium Agatston score >400.
* Diabetic men and women and two other risk factors
* Documented known CAD:
* Men and women asymptomatic or stable symptoms and known CAD by abnormal catheterization or prior SPECT without revascularization after >2 years to evaluate worsening disease or
* Men and women with worsening symptoms and known CAD by abnormal catheterization or prior SPECT/PET without revascularization
* Men and women with chest pain syndrome and previous revascularization
* Asymptomatic men and women >5 years after coronary artery bypass graft surgery (CABG) or >2 years after PCI

  * Risk factors: Diabetes, Current or recent cigarette smoking (within the last 12 months), LDL>130, low HDL <50 women, HDL <45 men, history of metabolic syndrome, hypertension (SPB>140), family history of premature (<60 year) CAD, Atherosclerotic carotid artery disease OR atherosclerotic peripheral vascular disease (APVD) as defined by ankle-brachial index below 0.9 and/or by abnormal duplex ultrasound, CT angiography, magnetic resonance angiography (MRA) or conventional invasive angiogram or previous revascularization procedure.

    * Framingham's high risk criteria refers to presence of diabetes mellitus with the limitation described above (c) or 10 year absolute Coronary Heart Disease(CHD)risk of >or= 20% (see tables Appendix A).

      * Chest pain is defined as Typical Angina if Exertional + Retrosternal + relieved with rest or sublingual nitroglycerin (NTG) , Atypical angina if only two of the above criteria are present and Non-anginal if one or none of the above are present.

Exclusion Criteria:

* Age <40
* Low pretest likelihood of CAD (= not meeting the above criteria)
* Unstable angina high risk (dynamic ST-Twave ECG changes and/or elevated troponin)
* Recent MI (<4 weeks)
* Recent stroke (<4 weeks)
* CABG or percutaneous coronary intervention (PCI) within the last 6 months
* Severe renal dysfunction as defined by creatinine > 2.0 mg/dl
* Active liver disease or hepatic dysfunction, AST or ALT > x 2 the upper limit of normal (ULN)
* Concomitant valvular heart disease
* Left ventricular ejection fraction (LVEF) <30%
* Severe systemic hypertension defined as systolic blood pressure (SBP) > 200 mmHg
* Symptomatic sustained or non-sustained ventricular tachycardia
* Morbid Obesity defined by Body Mass Index > 35
* Sever disability to prevent therapeutic exercise not expected to resolve within 6 months
* Major non-cardiac co-morbidity limiting survival or social situation/condition that in the opinion of the investigator will preclude the patient from participation in the study follow-up.
* Concurrent or prior (within last 30 days) participation in other research studies using investigational drugs or devices.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1085 (Actual)
Dates: Start 2009-03-11 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
1.Clinical Endpoints- | 2 years, 5 years and 10 years
  Average Risk Score modification during 5 year follow-up and major cardiovascular clinical events of death and non-fatal myocardial infarction.

SECONDARY OUTCOMES:
2. Secondary outcome | 2 years, 5 years and 10 years
  These measures are major events consisting of death, non-fatal MI, stroke, and revascularization procedures.

OTHER OUTCOMES:
Comprehensive economic analysis | 2 years, 5 years and 10 years
  Will compare total cost and health outcomes of treating patients at risk or with established CAD

CONTACTS AND LOCATIONS:
Overall Officials: K. Lance Gould, MD, Principal Investigator — University of Texas Medical Health Science Center at Houston
Locations (1):
- Weatherhead PET Center, Memorial Hermann Hospital TMC, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gould KL, Johnson NP, Roby AE, Kirkeeide R, Haynie M, Nguyen T, Bui L, Patel MB, Kitkungvan D, Mendoza P, Lai D, Li R, Sdringola S, McPherson D, Narula J. Optimal medical care and coronary flow capacity-guided myocardial revascularization vs usual care for chronic coronary artery disease: the CENTURY trial. Eur Heart J. 2025 Sep 2;46(33):3273-3286. doi: 10.1093/eurheartj/ehaf356. PMID 40439159
- [Derived] Kitkungvan D, Johnson NP, Kirkeeide R, Haynie M, Carter C, Patel MB, Bui L, Madjid M, Mendoza P, Roby AE, Hood S, Zhu H, Lai D, Sdringola S, Gould KL. Design and rationale of the randomized trial of comprehensive lifestyle modification, optimal pharmacological treatment and utilizing PET imaging for quantifying and managing stable coronary artery disease (the CENTURY study). Am Heart J. 2021 Jul;237:135-146. doi: 10.1016/j.ahj.2021.03.012. Epub 2021 Mar 21. PMID 33762179
- See also: For more information about cardiac PET imaging — http://www.uth.tmc.edu/pet/